CLINICAL TRIAL: NCT00079079
Title: A Phase II Study of Cisplatin and Gemcitabine in Patients With Locally Advanced/Recurrent or Metastatic Malignant Salivary Gland Tumors
Brief Title: Cisplatin or Carboplatin Combined With Gemcitabine in Locally Advanced, Recurrent, or Metastatic Malignant Salivary Gland Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN4; CAN-NCIC-HN4 (Other: PDQ); LILLY-CAN-NCIC-HN4 (Other: LILLY); CDR0000353487 (Other: PDQ)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Head and Neck Cancer
Keywords: stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; salivary gland acinic cell tumor; salivary gland adenoid cystic carcinoma; salivary gland poorly differentiated carcinoma; high-grade salivary gland mucoepidermoid carcinoma; low-grade salivary gland mucoepidermoid carcinoma; salivary gland malignant mixed cell type tumor; salivary gland adenocarcinoma; salivary gland anaplastic carcinoma; salivary gland squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms | interventions — Carboplatin; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, carboplatin, and gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with either cisplatin or carboplatin works in treating patients with locally advanced, recurrent, or metastatic malignant salivary gland tumor (cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the activity of cisplatin or carboplatin in combination with gemcitabine, in terms of response rate, in patients with locally advanced, recurrent, or metastatic malignant salivary gland tumor.

Secondary

* Determine the complete response in patients treated with these regimens.
* Determine the duration of response in patients treated with these regimens.
* Determine the toxicity profile of these regimens in these patients.
* Determine the overall survival of patients treated with these regimens.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes on days 1 and 8. Patients also receive either cisplatin IV over 1 hour on day 2 OR carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks, every 3 months for 1 year, and then every 6 months thereafter until relapse.

PROJECTED ACCRUAL: A total of 11- 34 patients will be accrued for this study within 1.5-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant salivary gland tumor

  * All histological subtypes eligible
  * Locally advanced, recurrent, or metastatic disease
  * Considered incurable by radiotherapy or surgery
  * Low- to intermediate-grade mucoepidermoid tumor or acinic cell carcinoma allowed provided patients are symptomatic OR at imminent risk of developing symptoms attributable to metastatic disease
* Disease must meet 1 of the following criteria:

  * Metastatic disease that is chemonaïve
  * Metastatic disease that has progressed after a prior non-cisplatin/carboplatin/gemcitabine regimen
  * Local and/or distant recurrence after curative surgery and/or radiotherapy
  * Locally advanced disease not suitable for surgery or radiotherapy
* At least 1 site of unidimensionally measurable disease documented by 1 of the following:

  * At least 20 mm by X-ray, physical exam, or non-spiral CT scan
  * At least 10 mm by spiral CT scan
* No bone metastases as only site of measurable disease
* No known brain metastasis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST/ALT no greater than 3 times upper limit of normal

Renal

* Creatinine clearance at least 60 mL/min (for cisplatin) OR 30-59 mL/min (for carboplatin)

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious illness or medical condition that would preclude study participation
* No active uncontrolled infection
* No neurologic disorder or psychiatric illness that would preclude study compliance
* No other malignancy within the past 5 years except adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy for locally advanced, recurrent, or metastatic disease and recovered

  * Must have been a non-cisplatin/carboplatin/gemcitabine-containing regimen
* More than 12 months since prior adjuvant chemotherapy (including cisplatin/carboplatin-based regimens) and recovered
* No prior gemcitabine

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to only site of measurable disease unless there is documented disease progression after therapy

Surgery

* See Disease Characteristics
* At least 21 days since prior surgery and recovered

Other

* More than 30 days since prior anticancer therapy
* More than 30 days since prior investigational agents
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2003-10-27 (Actual); Primary Completion 2008-09-29 (Actual); Study Completion 2009-02-10 (Actual)

PRIMARY OUTCOMES:
Objective response measured by RECIST criteria after accrual of 11 evaluable patients

SECONDARY OUTCOMES:
Toxicity assessed by NCI CTC v2.0
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Lillian L. Siu, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (4):
- Canada (4):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laurie SA, Siu LL, Winquist E, Maksymiuk A, Harnett EL, Walsh W, Tu D, Parulekar WR. A phase 2 study of platinum and gemcitabine in patients with advanced salivary gland cancer: a trial of the NCIC Clinical Trials Group. Cancer. 2010 Jan 15;116(2):362-8. doi: 10.1002/cncr.24745. PMID 19924794